CLINICAL TRIAL: NCT03346655
Title: Brain Metastases in Norway - Improved Classification and Treatment. A Prospective Cohort Study
Brief Title: Brain Metastases in Norway - A Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Olav Erich Yri, MD, PhD, Postdoctoral research fellow, Oslo University Hospital
Other Study IDs: 2017/1358
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Brain Metastases
Keywords: Treatment
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim and primary outcome of this study will be a descriptive analysis of the current treatment practice of BM in Norway. Specifically, it may give answers to the following research questions:

* What is the true incidence of BM in Norway?
* How are patients with BM treated at present?
* Do treatments differ between hospitals?
* How do treatments impact quality of life of the patients?
* Which factors (treatment, tumor and host variables) can explain disease control, survival, symptom relief, and general functions?
* How can BM staging be improved?

ELIGIBILITY:
Inclusion Criteria:

* Verified cancer diagnosis of solid tumors (based on radiological, histological/cytological or operative evidence).
* Brain metastases verified by computer tomography (CT), contrast-enhanced magnetic resonance imaging (MRI), or surgical biopsies
* Age ≥ 18 years
* Able to comply with study procedures
* Able to provide written informed consent after information in Norwegian

Exclusion Criteria:

* Primary brain tumors
* Primary hematological malignancies (lymphomas, leukemias)
* Previous diagnosis and/or treatment of BM
* Unable to produce written informed consent after information in Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With previously or newly diagnosed cancer With radiologically proven brain metastases
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival after diagnosis of brain metastases | Time from diagnosis of brain metastases till death of any cause, assessed up to 12 months
  Calculation of the overall survival times for each patient enrolled

SECONDARY OUTCOMES:
Treatment offered to patients diagnosed with brain metastases | 3 years
  Description of treatment offered
Changes in patient reported symptoms and quality of life items through EORTC questionnaire QLQ PAL15 and submodule BN20 | Monthly up to 12 months after inclusion
  Description of changes in patient reported outcomes through standardized questionnaires.European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer Patients receiving palliative care (EORTC QLQ-C15-PAL), covers items such as pain, physical and emotional functioning. The QLQ-BN20 contains questions on 7 single-item symptom scales (headaches, seizures, drowsiness, hair loss, itchy skin, leg weakness, and bladder control), and 4 multi-item scales (future uncertainty, visual disorder, motor dysfunction, and communication deficit). Patient's scores are translated into a scale from 1-100. A change of 10 points in one item is considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Olav E Yri, MD, Principal Investigator — Post-doc
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided